CLINICAL TRIAL: NCT06491238
Title: Light vs. Moderate Intensity Exercise in Individuals With Myasthenia Gravis
Acronym: MG-Ex
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A24-169
Record Dates: First submitted 2024-06-21; First posted 2024-07-09 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Myasthenia Gravis
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Light intensity Exercise (Experimental): Aerobic intensity levels: Heart rate reserve (HRR) 30-39%, 9-11 Borg Rate of Perceived Exertion (RPE) Strength intensity levels: %One Repetition Max (1RM) 40-50%, OMNI RPE 1-4
  Interventions: Behavioral: Light Intensity Exercise
- Moderate intensity Exercise (Experimental): Aerobic intensity levels: HRR 40-59%, 12-13 Borg RPE Strength intensity levels: %1RM 60-80%, OMNI RPE 5-6
  Interventions: Behavioral: Moderate Intensity Exercise

INTERVENTIONS:
Behavioral: Light Intensity Exercise — 12 weeks light intensity strength and endurance NeuroWell exercise program, specifically developed for individuals with neurological disorders or injuries. Participants have the intensity goals descripted in the experimental arm.
  Arms: Light intensity Exercise
Behavioral: Moderate Intensity Exercise — 12 weeks moderate intensity strength and endurance NeuroWell exercise program, specifically developed for individuals with neurological disorders or injuries. Participants have the intensity goals descripted in the experimental arm.
  Arms: Moderate intensity Exercise

SUMMARY:
The overall purpose of this pilot study is to examine the feasibility, acceptability, and tolerability of light and moderate intensity exercise in adults with MGeffect of light vs. moderate intensity exercise on health outcomes. Participants will be enrolled into the NeuroWell exercise program, which is geared toward individuals with neurological disorders or injuries and led by Certified Exercise Physiologists (CEPs) at the HealthPartners Neuroscience Center. A total of 20 people with MG will be enrolled in this study and participate in a small group exercise program 3 times a week for 12 weeks. Participants will be randomized into two exercise groups: 1) Light intensity or 2) Moderate intensity. We hypothesize that light and moderate intensity exercise will be feasible, acceptable, and tolerable in adults with MG and that individuals in the light intensity exercise group will be able to achieve the same improvement in health outcomes as the moderate intensity group.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide and provision of signed and dated informed consent form.
* Age 18-80
* Diagnosis of generalized MG.
* On a stable MG prescription medication regimen for the last 3 months.

Exclusion Criteria:

* Non-English speaking
* Regular exercise participation within the month prior to study enrollment or any outside exercise participation during the study intervention period.
* Significant cognitive impairment of any etiology that would impact study participation.
* History of heart failure, chronic lung disease, angina or any other condition that causes unreasonable shortness of breath on exertion.
* History of any serious neurological, psychiatric, or substance use disorders that would impact study participation.
* Women who are currently pregnant or planning to become pregnant during the study.
* Any other medical conditions that could affect their ability to participate in exercise for the study duration (as determined by study investigators).
* Active participation or past participation ≤3 months in any other interventional research study.
* Unwilling to participate in all study related activities.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-09-16 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility of light and moderate intensity exercise | 12 weeks
  Percent of participants recruited of potential participants contacted. Range: [0-100]. Higher percentage indicates higher feasibility
Acceptability of light and moderate intensity exercise | 12 weeks
  Percent of participants who complete the program of participants who start the program. Range: [0-100]. Higher percentage indicates higher acceptability
Tolerability of light and moderate intensity exercise | 12 weeks
  Percent of classes participants complete during the course of the program. Range: [0-100]. Higher percentage indicates higher tolerability.

SECONDARY OUTCOMES:
Cardiovascular Test - 6-minute walk test | 12 weeks
  Pre-post change in distance a person can walk during the 6-minute walk test. Change = Post distance - pre distance. Larger positive difference in distance indicates a larger improvement in cardiovascular health from pre-post program.
Cardiovascular and Strength test | 12 weeks
  Pre-post change in time it takes a person to transfer from seated to standing position and then back to seated position 5 times. Change = Post time- pre time. Larger positive difference in time indicates a larger improvement in cardiovascular health and strength from pre-post program.
Strength Test - 1-RM Upper Limb | 12 weeks
  Pre-post change in weight that can be lifted during the 1-RM test. Change = Post 1-RM upper limb weight -pre 1-RM upper limb weight. Larger positive difference in weight lifted indicates a larger improvement in upper limb strength from pre-post program.
Strength Test - 1-RM Lower Limb | 12 weeks
  Pre-post change in weight that can be lifted during the 1-RM test. Change = Post 1-RM lower limb weight -pre 1-RM lower limb weight. Larger positive difference in weight lifted indicates a larger improvement in lower limb strength from pre-post program.

CONTACTS AND LOCATIONS:
Locations (1):
- HealthPartners Neuroscience Center, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided